CLINICAL TRIAL: NCT03392506
Title: A Control Study of Intrathoracic Lymph Node in NSCLC Staging by EBUS-TBNA-RTE and Radiography
Brief Title: EBUS-TBNA-RTE VS Radiography in Staging of NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director,Endoscopy Department,Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201702
Record Dates: First submitted 2017-11-29; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: CP-EBUS; EBUS-TBNA; Real time elasticity; Staging of lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBUS-TBNA-RTE (Experimental): Patients do CT、 PETCT examination and EBUS-TBNA-RTE
  Interventions: Device: EBUS-TBNA-RTE

INTERVENTIONS:
Device: EBUS-TBNA-RTE — Every patient will do CT、 PETCT and EBUS-TBNA-RTE.These three kind of examination will have their own result.The three methods of inspection will be compared by diagnostic rate

SUMMARY:
The purpose of this study is to make a qualitative and quantitative analysis of the intrathoracic lymph nodes by CP-EBUS elastography for the first time, and to make a benign and malignant diagnosis.

DETAILED DESCRIPTION:
The newly developed convex array can be used to identify the hardness of the lymph nodes and estimate the benign and malignant lymph nodes indirectly through the quantitative and visualized analysis of the elastic coefficient of the bronchus through the CP-EBUS elastography mode.

The purpose of this study is to make a qualitative and quantitative analysis of the intrathoracic lymph nodes by CP-EBUS elastography for the first time, and to make a benign and malignant diagnosis.

120cases will be enrolled.Compared with the commonly used methods to evaluate intrathoracic lymph node metastasis, the accuracy of chest CT and PET-CT were compared. The lymph node staging method and the final pathological gold standard of the three groups were compared, so as to verify the accuracy and clinical popularization of the bronchial ultrasound elastography mode.

ELIGIBILITY:
Inclusion Criteria:

1. Intrathoracic lymph node enlargement
2. EBUS-TBNA operation can be performed

Exclusion Criteria:

1. Unable to cooperate with the experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of EBUS-TBNA-RTE | 1year
  By comparison of the diagnostic accuracy of CT ,PET-CT and EBUS-TBNA-RTE

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China